CLINICAL TRIAL: NCT05034315
Title: Effects of Whole Egg Consumption on Inflammation, Mood, and Recovery in Collegiate Female Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-309
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole egg consumption (Experimental)
  Interventions: Other: Whole egg consumption
- No egg control (No Intervention)

INTERVENTIONS:
Other: Whole egg consumption — The participants in the whole egg group consumed two whole eggs immediately after exercise.
  Arms: Whole egg consumption

SUMMARY:
The objectives were to investigate the effects of whole egg consumption by collegiate female gymnasts on inflammatory markers, mood, and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Membership on the university gymnastics team

Exclusion Criteria:

* egg allergies, asthma, coronary artery disease, depression, diabetes, hypertension, migraines, cancer or cancer-related complications, or auto-immune disorder

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Serum C-reactive protein (CRP) | 8 months
Serum interleukin-6 (IL-6) | 8 months
Serum soluble interleukin-6 receptor (sIL-6R) | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States